CLINICAL TRIAL: NCT01701544
Title: Double Blind, Randomised, Single Centre, Crossover Pilot Trial of Bilateral Nucleus Basalis of Meynert Deep Brain Stimulation to Improve Cognitive Deficits in Patients With Parkinson's Disease.
Brief Title: Nucleus Basalis Deep Brain Stimulation for Thinking & Memory Problems in Parkinson's.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11/0516
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Dementia in Parkinson's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBM DBS Off (Sham Comparator): NBM DBS switched off
  Interventions: Device: NBM DBS
- NBM DBS On (Active Comparator): NBM DBS Switched On
  Interventions: Device: NBM DBS

INTERVENTIONS:
Device: NBM DBS — Deep Brain Stimulation targeting the Nucleus Basalis of Meynert

SUMMARY:
We will perform a pilot study to evaluate the effectiveness of human NBM DBS at improving cognitive deficits in PD patients referred and eligible for conventional DBS treatment for coexisting motor impairments. Six patients with PD with both motor fluctuations and cognitive impairments (including but not restricted to deficits in attention and working memory) will have bilateral electrodes implanted to ensure that superficial contacts lie in the conventional motor GPi target, while the deepest electrical contacts lie in the NBM- (see figure 1). We will place electrodes using our conventional image guided, stereotactic frame-based procedure currently used in patients at NHNN. Patients will be randomised into 2 groups in a crossover trial design to have 3 month periods of NBM stimulation switched on or switched off separated by a 1 month washout period, following which the patient will cross over to have the opposite condition for a further 3 months- see timeline. At the end of the crossover period, all patients will be invited for continued follow up with stimulation switched on and will have neuropsychological evaluations at 6 monthly intervals. Patients will be given the option of receiving additional conventional stimulation to the motor GPi, through the higher contacts of each electrode, at the end of the crossover period.

ELIGIBILITY:
Inclusion Criteria:

* All patients will meet Queen Square brain bank criteria for the diagnosis of PD and will have motor fluctuations (off periods and/or L-dopa induced dyskinesias) in response to medications that are known to improve with GPi DBS, and will be appropriate candidates for GPi DBS aside from the coexistence of cognitive impairment.

Patients will be aged between 35 and 80 years.

Patients will be able to give informed consent.

Patients will meet criteria for PD dementia. Patients will have a MMSE score between 26 and lower cutoff of 21 to restrict the sample to those with mild dementia and cognitive impairment. This will be equivalent to an age and education adjusted scaled score of greater than 5 and lower than 9 (mildly impaired range) on the Mattis Dementia Rating Scale-2.

Patients will have only minimal atrophy on pre-operative brain MRI scans.

Patients will be living at home and will have a carer living with them e.g. their spouse

Able to comply with trial protocol and willing to attend clinic necessary visits

Exclusion Criteria:

* Diagnosis or suspicion of other cause for parkinsonism or dementia.

Known abnormality on CT or MRI brain imaging considered likely to compromise compliance with trial protocol.

Prior intra-cerebral surgical intervention for Parkinson's disease including Deep Brain stimulation, lesional surgery, growth factor administration, gene therapy or cell transplant.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Abbreviated cognitive battery | 6 months
  Differences between each item of the abbreviated cognitive battery scores between patients after 3 months ON stimulation and 3 months OFF stimulation.
  CVLT-II,Verbal Fluency,Simple & Choice RT (CANTAB),Digit span,Posner's covert attention test

SECONDARY OUTCOMES:
Minimental State Examination | 6 months
DRS-2 | 6 months
  Dementia Rating Scale-2
SRM (Faces) | 6 months
  Short Recognition Memory for faces
WAIS-III (Letter number sequencing, Arithmetic) | 6 months
  Wechsler Abbreviated Scale of Intelligence
FAST | 6 months
  Florida Apraxia Screening test
NPI | 6 months
  Neuropsychiatric Inventory
BDS | 6 months
  Blessed Dementia Scale
HAM-D | 6 months
  Hamilton Depression scale
MDS UPDRS | 6 months
  Movement Disorders Society - Unified Parkinson's disease Rating scale
PDQ39 | 6 months
  Parkinson's disease quality of life questionnaire
GFQ | 6 months
  Gait and falls questioannaire
NMS Quest | 6 months
  Non Motor Symptoms Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Foltynie, PhD, Principal Investigator — UCL Institute of Neurology
Locations (1):
- National Hospital for Neurology & Neurosurgery, London, United Kingdom

REFERENCES:
- [Derived] Gratwicke J, Zrinzo L, Kahan J, Peters A, Beigi M, Akram H, Hyam J, Oswal A, Day B, Mancini L, Thornton J, Yousry T, Limousin P, Hariz M, Jahanshahi M, Foltynie T. Bilateral Deep Brain Stimulation of the Nucleus Basalis of Meynert for Parkinson Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):169-178. doi: 10.1001/jamaneurol.2017.3762. PMID 29255885